CLINICAL TRIAL: NCT05454553
Title: Efficacity of Deep Inspiration Breath Hold and Intensity-modulated Radiotherapy in Preventing PErfusion Defect for Left Sided Breast Cancer (EDIPE)
Acronym: EDIPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-012; ID-RCB (Other: 2022-A00320-43)
Record Dates: First submitted 2022-06-22; First posted 2022-07-12 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cardiac Toxicity; Deep Inspiration Breath Hold; Myocardial Perfusion Imaging
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with left sided breast cancer who are planned for (Experimental): one of the following heart sparing techniques :
  * DIBH radiotherapy
  * IMRT
  Interventions: Other: myocardial perfusion SPECT

INTERVENTIONS:
Other: myocardial perfusion SPECT — For all participants, myocardial perfusion SPECT will be performed :
  at 3, 6 and 12 months (post irradiation)

SUMMARY:
Breast irradiation is known to cause radiation-induced heart disease (RIHD) many years later after radiotherapy. Recent studies suggest that RIHD could be an earlier complication and that subclinical cardiac injury can be detected such as myocardial perfusion defects. Myocardial perfusion single photon emission computed tomography (SPECT) is a sensitive and specific technique able to detect perfusion abnormalities which are more frequent in left-sided breast cancer patients because of the cardiac exposure.

The most used technique for breast cancer irradiation is tangential opposed field, but this technique exposes the left anterior descending coronary artery to high dose during left breast irradiation.

There are different cardiac sparing techniques to reduce heart exposure such as:

* Deep inspiration breath-hold (DIBH) which displaces the heart out of the radiation beam
* Intensity-modulated radiation therapy (IMRT) which decreases heart exposure to high doses but changes the dose distribution in the heart and increases lower doses.

DETAILED DESCRIPTION:
In breast radiotherapy, especially for left sides breast cancers, the heart is the organ-at-risk which whose dose constraints are source of controversies. Historically breast cancer radiation therapy was associated with a significantly increased cardiac mortality. Two meta-analyses founded that the cardiac mortality risk was increased by 27% to 38%. This result is linked to outdated 2-D treatment techniques causing massive cardiac overexposure (Clarke M et al. 2005, Cheng YJ et al. 2017).

Three dimensional conformational radiotherapy reduced mean heart dose but the link between heart irradiation and radiation-induced heart damages doesn't seem to have threshold therefore to RHID is still a matter of concern (Darby SC et al. 2013; Taylor C et al. 2017).

The most used technique for breast cancer irradiation is opposite tangential field radiotherapy, however, it exposes the anterior interventricular coronary artery to a high dose during left breast irradiation (Nieder C et al. 2007). Therefore, radiotherapy techniques have developed to reduce cardiac exposure such as deep inspiration breath hold (DBIH) and intensity modulated radiation therapy (IMRT).

DBIH "mechanically" moves the heart away from the radiation beam and IMRT the dose distribution in the heart and reduces its exposure to high doses (Boda-Heggemann J et al. 2016, Lauche O et al. 2016).

Nevertheless, recent studies suggest that even with this level of cardiac exposure subclinical cardiac alterations may be detected, such as myocardial perfusion deficit (Eber et al. 2022; Marks LB et al. 2005; Gyenes G et al. 1997; Sioka C et al. 2011; Seddon B et al. 2002; Eftekhari M et al. 2015).

The heart is a complex and heterogeneous organ, however it's mostly considered as an homogeneous organ-at-risk during treatment planning in daily practice. Dosimetric optimization is therefore mainly performed on the global cardiac structure and the mean cardiac dose (MHD). Dosimetric studies reported a poor correlation between MHD and mean doses to cardiac substructures questioning the relevance of the MHD as a reflection of the dose distribution to the heart (Jacob S et al. 2016).

Recent data suggested to take account of the histological diversity and the functional complexity of the cardiac substructure (Darby SC et al. 2010; Gillette EL et al. 1985; Ghita M et al. 2020; Eber J et al. 2021). This delineation is not performed in routine clinical practice due to the poorly reproducible and time-consuming manual contouring.

The development of auto-segmentation software can save time and improve the quality of the delineation process of these substructures in order to optimize dosimetry (Feng M et al. 2011; Maffei N et al. 2020).

The investigators propose a single-centre prospective study to evaluate the utility of deep inspiration breath hold using a surface monitoring technique (AlignRT, Vision RT Ltd., London, UK) and IMRT, as means to prevent the development of myocardial perfusional deficits in patients treated for left breast cancer, using stress and, if necessary, resting myocardial scintigraphy.

Before initiation of radiotherapy patients will performed a chest CT scan in the treatment position for 3D treatment planning and dose calculation; a chest CT angiography for delineation of cardiac substructures; and a myocardial perfusion SPECT imaging to provide a map of regional myocardial perfusion and determine left ventricle ejection fraction (LVEF).

Treatment phase will consist of the standard course of breast radiotherapy in our department. The main difference will be in the delineation of the organ at risk, cardiac substructures will be delineated to obtain the dosimetry During the follow up period, patient will be scheduled to undergo cardiac SPECT before and at 3-, 6-, and 12-month period post irradiation. Stress ECG-gated SPECT will be performed after infusion of 3 MBq/kg 99mTc-tetrofosmin (Myoview®, General Electrics Healthcare) at peak pharmacological stress with regadenoson, (single dosage: 400 µg; Rapiscan®, GE healthcare)

ELIGIBILITY:
Inclusion Criteria:

* Patient with left sided breast cancer histologically confirmed after lumpectomy or mastectomy with/without lymph node involvement who are planned for DIBH-RT or IMRT
* Age > 18 years
* Karnofsky Performance Status (KPS) > 60%
* Absence of psychiatric illness hindering follow-up
* Patient understands French
* Signature of informed consent
* Patient registered with social security

Exclusion Criteria:

* Bilateral breast cancer
* History of thoracic irradiation
* Pregnancy or breastfeeding
* Any medical contraindication of cardiac SPECT or chest CT angiography.
* Any medical contraindication of Regadenoson

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-10-27 (Estimated); Study Completion 2024-10-27 (Estimated)

PRIMARY OUTCOMES:
Evaluation of DIBH and IMRT efficacy in preventing perfusion defect for left-sided breast cancer after radiotherapy | at 3 months from the end of radiotherapy
  Incidence of perfusion defects on follow-up myocardial perfusion SPECT scans
Evaluation of DIBH and IMRT efficacy in preventing perfusion defect for left-sided breast cancer after radiotherapy | at 6 months from the end of radiotherapy
  Incidence of perfusion defects on follow-up myocardial perfusion SPECT scans
Evaluation of DIBH and IMRT efficacy in preventing perfusion defect for left-sided breast cancer after radiotherapy | at 12 months from the end of radiotherapy
  Incidence of perfusion defects on follow-up myocardial perfusion SPECT scans

SECONDARY OUTCOMES:
Assession of wall-motion abnormalities and left ventricular ejection fraction (LVEF) decrease | up to 12 months from the end of radiotherapy
  Incidence of left ventricular wall motion disorder and LVEF quantification on follow-up myocardial perfusion SPECT scans.
Assessing the relevance of mean heart dose in the prevention of Radiation-induced heart disease (RIHD) compared to cardiac substructures. | up to 12 months from the end of radiotherapy
  Measurement of the doses delivered to the cardiac volumes and its substructures.
Influence of cardiac risk factors on post-radiation myocardial perfusion. | up to 12 months from the end of radiotherapy
Influence of anticancer therapy exposure on post-radiation myocardial perfusion | up to 12 months from the end of radiotherapy
  Anticancer therapy characteristics (type)
Influence of anticancer therapy exposure on post-radiation myocardial perfusion | up to 12 months from the end of radiotherapy
  Anticancer therapy characteristics (dose)
Influence of anticancer therapy exposure on post-radiation myocardial perfusion | up to 12 months from the end of radiotherapy
  Anticancer therapy characteristics (duration)
Impact of the location of the tumor bed boost on the cardiac dose. | up to 12 months from the end of radiotherapy
  Location of the tumor bed boost
Impact of the location of the tumor bed boost on the cardiac dose. | up to 12 months from the end of radiotherapy
  Cardiac dose

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France

REFERENCES:
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Cheng YJ, Nie XY, Ji CC, Lin XX, Liu LJ, Chen XM, Yao H, Wu SH. Long-Term Cardiovascular Risk After Radiotherapy in Women With Breast Cancer. J Am Heart Assoc. 2017 May 21;6(5):e005633. doi: 10.1161/JAHA.117.005633. PMID 28529208
- [Background] Darby SC, Ewertz M, McGale P, Bennet AM, Blom-Goldman U, Bronnum D, Correa C, Cutter D, Gagliardi G, Gigante B, Jensen MB, Nisbet A, Peto R, Rahimi K, Taylor C, Hall P. Risk of ischemic heart disease in women after radiotherapy for breast cancer. N Engl J Med. 2013 Mar 14;368(11):987-98. doi: 10.1056/NEJMoa1209825. PMID 23484825
- [Background] Taylor C, Correa C, Duane FK, Aznar MC, Anderson SJ, Bergh J, Dodwell D, Ewertz M, Gray R, Jagsi R, Pierce L, Pritchard KI, Swain S, Wang Z, Wang Y, Whelan T, Peto R, McGale P; Early Breast Cancer Trialists' Collaborative Group. Estimating the Risks of Breast Cancer Radiotherapy: Evidence From Modern Radiation Doses to the Lungs and Heart and From Previous Randomized Trials. J Clin Oncol. 2017 May 20;35(15):1641-1649. doi: 10.1200/JCO.2016.72.0722. Epub 2017 Mar 20. PMID 28319436
- [Background] Nieder C, Schill S, Kneschaurek P, Molls M. Influence of different treatment techniques on radiation dose to the LAD coronary artery. Radiat Oncol. 2007 Jun 5;2:20. doi: 10.1186/1748-717X-2-20. PMID 17547777
- [Background] Boda-Heggemann J, Knopf AC, Simeonova-Chergou A, Wertz H, Stieler F, Jahnke A, Jahnke L, Fleckenstein J, Vogel L, Arns A, Blessing M, Wenz F, Lohr F. Deep Inspiration Breath Hold-Based Radiation Therapy: A Clinical Review. Int J Radiat Oncol Biol Phys. 2016 Mar 1;94(3):478-92. doi: 10.1016/j.ijrobp.2015.11.049. Epub 2015 Dec 17. PMID 26867877
- [Background] Lauche O, Kirova YM, Fenoglietto P, Costa E, Lemanski C, Bourgier C, Riou O, Tiberi D, Campana F, Fourquet A, Azria D. Helical tomotherapy and volumetric modulated arc therapy: New therapeutic arms in the breast cancer radiotherapy. World J Radiol. 2016 Aug 28;8(8):735-42. doi: 10.4329/wjr.v8.i8.735. PMID 27648167
- [Background] Eber J, Leroy-Freschini B, Antoni D, Noel G, Pflumio C. Increased cardiac uptake of (18F)-fluorodeoxyglucose incidentally detected on positron emission tomography after left breast irradiation: How to interpret? Cancer Radiother. 2022 Sep;26(5):724-729. doi: 10.1016/j.canrad.2021.10.010. Epub 2022 Feb 12. PMID 35165015
- [Background] Marks LB, Yu X, Prosnitz RG, Zhou SM, Hardenbergh PH, Blazing M, Hollis D, Lind P, Tisch A, Wong TZ, Borges-Neto S. The incidence and functional consequences of RT-associated cardiac perfusion defects. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):214-23. doi: 10.1016/j.ijrobp.2005.01.029. PMID 16111592
- [Background] Gyenes G, Fornander T, Carlens P, Glas U, Rutqvist LE. Detection of radiation-induced myocardial damage by technetium-99m sestamibi scintigraphy. Eur J Nucl Med. 1997 Mar;24(3):286-92. doi: 10.1007/BF01728765. PMID 9143466
- [Background] Sioka C, Exarchopoulos T, Tasiou I, Tzima E, Fotou N, Capizzello A, Ragos V, Tsekeris P, Fotopoulos A. Myocardial perfusion imaging with (99 m)Tc-tetrofosmin SPECT in breast cancer patients that received postoperative radiotherapy: a case-control study. Radiat Oncol. 2011 Nov 8;6:151. doi: 10.1186/1748-717X-6-151. PMID 22067743
- [Background] Seddon B, Cook A, Gothard L, Salmon E, Latus K, Underwood SR, Yarnold J. Detection of defects in myocardial perfusion imaging in patients with early breast cancer treated with radiotherapy. Radiother Oncol. 2002 Jul;64(1):53-63. doi: 10.1016/s0167-8140(02)00133-0. PMID 12208576
- [Background] Eftekhari M, Anbiaei R, Zamani H, Fallahi B, Beiki D, Ameri A, Emami-Ardekani A, Fard-Esfahani A, Gholamrezanezhad A, Seid Ratki KR, Roknabadi AM. Radiation-induced myocardial perfusion abnormalities in breast cancer patients following external beam radiation therapy. Asia Ocean J Nucl Med Biol. 2015 Winter;3(1):3-9. PMID 27408875
- [Background] Jacob S, Pathak A, Franck D, Latorzeff I, Jimenez G, Fondard O, Lapeyre M, Colombier D, Bruguiere E, Lairez O, Fontenel B, Milliat F, Tamarat R, Broggio D, Derreumaux S, Ducassou M, Ferrieres J, Laurier D, Benderitter M, Bernier MO. Early detection and prediction of cardiotoxicity after radiation therapy for breast cancer: the BACCARAT prospective cohort study. Radiat Oncol. 2016 Apr 7;11:54. doi: 10.1186/s13014-016-0627-5. PMID 27056179
- [Background] Darby SC, Cutter DJ, Boerma M, Constine LS, Fajardo LF, Kodama K, Mabuchi K, Marks LB, Mettler FA, Pierce LJ, Trott KR, Yeh ET, Shore RE. Radiation-related heart disease: current knowledge and future prospects. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):656-65. doi: 10.1016/j.ijrobp.2009.09.064. PMID 20159360
- [Background] Gillette EL, McChesney SL, Hoopes PJ. Isoeffect curves for radiation-induced cardiomyopathy in the dog. Int J Radiat Oncol Biol Phys. 1985 Dec;11(12):2091-7. doi: 10.1016/0360-3016(85)90089-6. PMID 4066441
- [Background] Ghita M, Gill EK, Walls GM, Edgar KS, McMahon SJ, Osorio EV, Bergom C, Grieve DJ, Watson CJ, McWilliam A, Aznar M, van Herk M, Williams KJ, Butterworth KT. Cardiac sub-volume targeting demonstrates regional radiosensitivity in the mouse heart. Radiother Oncol. 2020 Nov;152:216-221. doi: 10.1016/j.radonc.2020.07.016. Epub 2020 Jul 12. PMID 32663535
- [Background] Eber J, Nannini S, Chambrelant I, Le Fevre C, Noel G, Antoni D. [Impact of thoracic irradiation on cardiac structures]. Cancer Radiother. 2022 May;26(3):526-536. doi: 10.1016/j.canrad.2021.08.022. Epub 2021 Oct 30. French. PMID 34728116
- [Background] Feng M, Moran JM, Koelling T, Chughtai A, Chan JL, Freedman L, Hayman JA, Jagsi R, Jolly S, Larouere J, Soriano J, Marsh R, Pierce LJ. Development and validation of a heart atlas to study cardiac exposure to radiation following treatment for breast cancer. Int J Radiat Oncol Biol Phys. 2011 Jan 1;79(1):10-8. doi: 10.1016/j.ijrobp.2009.10.058. Epub 2010 Apr 24. PMID 20421148
- [Background] Maffei N, Fiorini L, Aluisio G, D'Angelo E, Ferrazza P, Vanoni V, Lohr F, Meduri B, Guidi G. Hierarchical clustering applied to automatic atlas based segmentation of 25 cardiac sub-structures. Phys Med. 2020 Jan;69:70-80. doi: 10.1016/j.ejmp.2019.12.001. Epub 2019 Dec 10. PMID 31835189